CLINICAL TRIAL: NCT03630796
Title: Effect of Sevoflurane Anesthesia in Postoperative Troponin I Levels in Children Undergoing Congenital Heart Defects Surgery: a Randomized Controlled Clinical Trial
Brief Title: Effect of Sevoflurane in Postoperative Troponin I Levels in Children Undergoing Congenital Heart Defects Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto do Coracao (Other Government)
Responsible Party: Principal Investigator, Filomena R B G Galas, Phd MD, Instituto do Coracao
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4343.19.009
Record Dates: First submitted 2018-08-10; First posted 2018-08-15 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Congenital Heart Defects
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Sevoflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sevoflurane (Active Comparator): Anesthetic induction with sevoflurane by mask 3-8% and fresh gas flow 2-8 l/min (FiO2 50-100%) followed by ketamine 1-2 mg/kg, midazolam 0,1-0,5 mg/kg, fentanyl 2-4 mcg/kg and pancuronium 0,1 mg/kg.
  After orotracheal intubation, anesthesia is maintained with fentanyl 10 - 30 mcg/kg according to clinical needs and sevoflurane 1-3% (end-tidal concentration) before and after cardiopulmonary bypass. Specifically during cardiopulmonary bypass extra fentanyl 1-5 mcg/kg and pancuronium 0,1 mg/kg will be administered and the sevoflurane sustained 1-3% in a specific sevoflurane vaporizer included in the CPB machine.
  Pressure-controlled ventilation will be applied to both groups objectifying normocarbia and normoxia.
  Ringer's lactate (RL) will be used as crystalloid solution for fluid therapy.
  Interventions: Drug: Sevoflurane
- Intravenous anesthetics (TIVA) (Other): Anesthetic induction with ketamine 1-3 mg/kg, midazolam 0,1-0,5 mg/kg, fentanyl 2-4 mcg/kg and pancuronium 0,1 mg/kg after preoxygenation with FiO2 between 50-100% and fresh gas flow 4-8 l/min.
  After orotracheal intubation, anesthesia is maintained with fentanyl 10 - 30 mcg/kg according to clinical needs and continuous infusion of midazolam and ketamine 0,2-0,8 mg/kg/h and 1-2 mg/kg/h respectively before and after cardiopulmonary bypass. Specifically during cardiopulmonary bypass extra fentanyl 1-5 mcg/kg, midazolam 0,1-0,5 mg/kg and pancuronium 0,1 mg/kg will be administered.
  Pressure-controlled ventilation will be applied to both groups objectifying normocarbia and normoxia.
  Ringer's lactate (RL) will be used as crystalloid solution for fluid therapy.
  Interventions: Drug: TIVA

INTERVENTIONS:
Drug: Sevoflurane — Use of sevoflurane (compared to total intravenous anesthesia) in congenital heart deffects surgeries.
  Arms: Sevoflurane
Drug: TIVA — Total intravenous anesthesia
  Arms: Intravenous anesthetics (TIVA)

SUMMARY:
The main purpose of this study is to compare myocardial injury of patients undergoing congenital cardiac defects repair surgery (RACHS Risk Score one, two or three) under total intravenous anesthesia compared to inhalation anesthesia with sevoflurane. The primary aim of the study is to evaluate the troponin I levels in patients following congenital heart surgery and elucidate if one of the two anesthetic techniques (TIVA x inhalation anesthesia) is more effective in reducing troponin I levels in the first 72h after surgery..

Sixty six are planned to be included in the study and the follow-up will take approximately 3 days for the primary outcome.

As a secondary outcome evaluate the BNP, CPK and CKMB postoperative levels in the same period (72h), also ICU and hospital lengh of stay (LOS), duration of mechanical ventilation, inotropic/vasoactive drugs use and incidence of renal injury (according to pediatric RIFLE score).

ELIGIBILITY:
Inclusion Criteria

* Written informed consent (signed by the parents)
* Scheduled Congenital Heart Defect Repair Surgery RACHS Risk Score 1, 2 or 3. On-pump Surgery
* Age: 2 years old (completed) or younger
* Patients without previous kidney disease or any contraindication for inhaled anesthesia (including previous unusual response to an anesthetic agent)
* No previous general anesthesia in the last 30 days.

Exclusion Criteria

* Emergency surgery
* Off-pump surgery (surgery plan changed by the surgeon after patient's randomization)
* Refuse to take part of the study or ask to leave the trial

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2018-08-20 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Serum levels curve of troponin I | T0: induction anesthesia; T1: ICU admission; T2: 24 hours after surgery; T3: 48 hours after surgery; T4: 72 hours after surgery
  Dosage of serum troponin I during the first 72 hours after surgery

SECONDARY OUTCOMES:
Serum levels curve of CKMB, CPK and BNP | T0: induction anesthesia; T1: ICU admission; T2: 24 hours after surgery; T3: 48 hours after surgery; T4: 72 hours after surgery
  Dosage of serum CKMB, CPK and BNP during the first 72 hours after surgery
Acute kidney injury | within 30 days after cardiac surgery
  According to pediatric RIFLE
Cardiac complications | within 30 days after cardiac surgery
  Arrhythmia, low cardiac output syndrome
Blood transfusion | within 30 days after cardiac surgery
Length of vasoactive drugs | within 30 days after cardiac surgery
Duration of Mechanical ventilation | within 30 days after cardiac surgery
Length of ICU stay | within 30 days after cardiac surgery
Length of hospital stay | within 30 days after cardiac surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Incor - Heart Institute - University of Sao Paulo, São Paulo, Brazil